CLINICAL TRIAL: NCT01598987
Title: A 24-month, Multi-center, Single Arm, Prospective Study to Evaluate Renal Function, Efficacy, Safety and Tolerability of Everolimus in Combination With Reduced Exposure Cyclosporine or Tacrolimus in Paediatric Liver Transplant Recipients.
Brief Title: Efficacy, Safety and Tolerability of Everolimus in Combination With Reduced Exposure Cyclosporine or Tacrolimus in Paediatric Liver Transplant Recipients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001H2305; 2011-003069-14
Record Dates: First submitted 2012-03-01; First posted 2012-05-15 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Renal Function; Liver Transplant
Keywords: Paediatric liver transplantation; Everolimus; Reduced calcineurin inhibitor; Cyclosporine, tacrolimus; Renal function; Composite efficacy endpoint (treated biopsy proven acute rejection death, graft loss); Liver transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus based regimen (Experimental): Conversion at Baseline from an immunosuppressive regimen which contains either cyclosporine (CsA) or tacrolimus (TAC) with or without mycophenolic acid (MPA), with or without corticosteroids in a regimen which contains everolimus combined reduced dose of either cyclosporine (CsA) or tacrolimus (TAC).
  The dosing schedule was twice daily, 12 hours apart.
  Interventions: Drug: Introduction of everolimus with reduced cyclosporine or tacrolimus dose, the earliest 1 month and the latest 6 months after liver transplantation.

INTERVENTIONS:
Drug: Introduction of everolimus with reduced cyclosporine or tacrolimus dose, the earliest 1 month and the latest 6 months after liver transplantation. — Immunosuppression after liver transplantation. Pediatric transplant recipients received a starting dose of 0.8 mg/m^2/dose in combination wit Cyclosporine A or 2.0 mg/m^2/dose in combination with tacrolimus, twice-daily. Thereafter, doses were adjusted to achieve everolimus C-0h blood trough level between 3 to 8 ng/ml.

SUMMARY:
This study was designed to assess the evolution of renal function and to collect efficacy, safety, and tolerability data of everolimus in co-exposure with reduced CNI in paediatric liver transplant recipients.

DETAILED DESCRIPTION:
Study is completed (was active and ongoing but no longer recruiting since December 2014). The study Data Monitoring Committee meeting communicated to Novartis the following safety findings in the study population: high rate of premature discontinuation of study medication, high rate of post-transplant lymphoproliferative disease and high rate of related serious infections leading to hospitalization. In light of the safety findings, Novartis followed the DMC recommendation to discontinue the study medication in this age group and to stop enrolling new patients in this study (regardless of age).

ELIGIBILITY:
Key Inclusion Criteria:

Signed informed consent from both parents or legal guardian(s) prior to patient participation in the study.

Paediatric liver transplant recipients aged greater than or equal to 1 month and younger than 18 years of age.

Paediatric recipients at the earliest 1 month and latest 6 month after liver transplantation.

Key Exclusion Criteria:

Patients with hepato-biliary malignancies and/or patients transplanted due to fulminant hepatitis /acute liver failure.

Presence of thrombosis of any major hepatic arteries, major/reconstructed hepatic veins, portal vein or inferior vena cava at any time prior to the start of study drug.

Patients with serum creatinine value >2 times age-related ULN at Baseline or who received renal replacement therapy within one week prior to the start of study drug and patients with a confirmed spot urine protein/creatinine ratio indicating a urinary protein excretion >500 mg/m2/24 hrs, at Baseline.

Patients with clinically significant systemic infection and/or in a critical care setting requiring life support measures such as mechanical ventilation, dialysis, or vasopressor agents.

Patients with a known hypersensitivity to the drugs used on study or their class, or to any of the excipients.

Pregnant or nursing (lactating) female patients, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive βHCG laboratory test (>9 mIU/mL) at Baseline.

Female patients of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they agree for abstinence from sexual activity.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (31):
- United States (9):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Madison, Wisconsin
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Edmonton, Alberta, Canada
- Novartis Investigative Site, København Ø, Denmark
- Novartis Investigative Site, Bron, France
- Germany (6):
  - Novartis Investigative Site, Hanover, Germany
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Budapest, Hungary
- Italy (4):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Roma, ITA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Torino, TO
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Stockholm, Sweden
- United Kingdom (3):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 62 patients were screened prior to the data monitoring committee (DMC) recommendation to terminate enrolment.
  Six patients were screen failures. The other 56 patients were included and treated.
Groups:
- Everolimus Based Regimen: Conversion at baseline from an immunosuppressive regimen which contains either cyclosporine (CsA) or tacrolimus (TAC) with or without mycophenolic acid (MPA), with or without corticosteroids to a regimen which contains everolimus combined with reduced dose of either cyclosporine (CsA) or tacrolimus (TAC).
  The dosing schedule was twice daily, 12 hours apart.
Period: Baseline to Month 12
Arm/Group | Everolimus Based Regimen
Started | 56
Completed | 50
Not Completed | 6
Not completed — Administrative problems | 2
Not completed — Withdrawal by Subject | 4
Period: Baseline to 24 Month
Arm/Group | Everolimus Based Regimen
Started | 56
Completed | 48
Not Completed | 8
Not completed — Withdrawal by Subject | 5
Not completed — Administrative problems | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): consisted of all patients enrolled into the study, including patients who did not receive any everolimus, but were followed beyond baseline.
Arm/Group | Everolimus Based Regimen
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.9 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate - Month 12
Description: Evolution of renal function assessed by estimated Glomerular Filtration Rate (eGFR) calculated by the Chronic Kidney Disease in Children (CKiD) Schwartz formula (Schwartz 2009), expressed in mean change in eGFR of CKiD between start of study (baseline assessment) and Month 12.
Time Frame: Baseline, Month 12
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Everolimus Based Regimen
Number analyzed (Participants) | 50
mL/min/1.73m^2 | 6.2 (19.52)

2. Secondary Outcome: Kaplan-Meier Estimates for Failure Rates of Efficacy Endpoints
Description: The proportion of patients with composite efficacy failure (treated biopsy proven acute rejection[tBPAR], graft loss [GL] , death [D]) before/at Month 12 and Month 24, estimated with Kaplan-Meier (KM) methods and the proportion of patients who experienced any of the components of composite efficacy failure (tBPAR, GL, D) before/at Month 12 and Month 24, separately for each component.
  AR: acute rejection; BPAR: biopsy proven acute rejection. Rate = Kaplan-Meier estimate for failure in %; CI = confidence interval for failure rate.
Time Frame: At 12-month and 24-month after start of study drug
Population: Full Analysis Set
Measure: Number (80% Confidence Interval); unit: Percentages
Arm/Group | Everolimus Based Regimen
Number analyzed (Participants) | 56
Percentages
  Month 12: tBPAR,GL,or D | 1.9 [0.0 to 4.2]
  Month 12: tBPAR,GL,D,or loss to follow-up | 1.9 [0.0 to 4.2]
  Month 12: Treated BPAR | 1.9 [0.0 to 4.2]
  Month 12: Graft loss | 0.0 [0.0 to 0.0]
  Month 12: Death | 0.0 [0.0 to 0.0]
  Month 12: Graft loss or death | 0.0 [0.0 to 0.0]
  Month 12: BPAR | 3.7 [0.4 to 7.0]
  Month 12: Treated AR | 3.6 [0.4 to 6.9]
  Month 24: tBPAR,GL,or D | 5.9 [0.3 to 11.5]
  Month 24: tBPAR,GL,D,or loss to follow-up | 9.7 [2.5 to 16.9]
  Month 24: Treated BPAR | 5.9 [0.3 to 11.5]
  Month 24: Graft Loss | 0.0 [0.0 to 0.0]
  Month 24: Death | 0.0 [0.0 to 0.0]
  Month 24: Graft loss or death | 0.0 [0.0 to 0.0]
  Month 24: BPAR | 11.9 [4.2 to 19.6]
  Month 24: Treated AR | 7.7 [1.7 to 13.6]

3. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate - Month 24
Description: Evolution of renal function assessed by estimated Glomerular Filtration Rate (eGFR) calculated by the Chronic Kidney Disease in Children (CKiD) Schwartz formula (Schwartz 2009), expressed in mean change in eGFR of CKiD between start of study (baseline assessment) and Month 24.
Time Frame: Baseline, Month 24
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Everolimus Based Regimen
Number analyzed (Participants) | 50
mL/min/1.73m2 | 4.5 (19.55)

4. Secondary Outcome: Growth Development - Height at Baseline and Month 12
Description: Individual growth measurements were compared with the gender and age-specific growth percentiles in the CDC growth charts for the US population. Each value observed is thus represented by the (approximated) percentage of subjects with a lower value in the reference population. Changes were calculated on this scale and thus express the change in growth measurements relative to the percentiles in the CDC growth charts.
  Patients were classified into growth percentile categories (<=5, >5-25, >25-50, >50-75, >75-95 and >95% percentile).
Time Frame: Baseline, Month 12
Population: Safety Analysis Set
Measure: Number; unit: Percentages
Groups:
- <=5% Percentile; >5% - 25% Percentile; >25% - 50% Percentile; >75% - 95% Percentile; >95% Percentile: Growth percentile category
- >50% - 75% Percentile: Growth percentile categpru
- Total: The classified change from baseline in growth percentiles cross-tabulated against baseline categories of growth percentiles.
Arm/Group | <=5% Percentile | >5% - 25% Percentile | >25% - 50% Percentile | >50% - 75% Percentile | >75% - 95% Percentile | >95% Percentile | Total
Number analyzed (Participants) | 16 | 15 | 6 | 7 | 4 | 2 | 50
Percentages
  Decrease | 0.0 | 26.7 | 16.7 | 14.3 | 25.0 | 0.0 | 14.0
  No Change | 68.8 | 20.0 | 33.3 | 28.6 | 50.0 | 100.0 | 44.0
  Increase >3 to 5% | 12.5 | 6.7 | 0.0 | 0.0 | 25.0 | 0.0 | 8.0
  Increase >5 to 10% | 0.0 | 20.0 | 16.7 | 14.3 | 0.0 | 0.0 | 10.0
  Increase >10% | 18.8 | 26.7 | 33.3 | 42.9 | 0.0 | 0.0 | 24.0

5. Secondary Outcome: Growth Development - Weight at Baseline and Month 12
Description: as for outcome 4
Time Frame: Baseline, Month 12
Population: Safety Analysis Set
Measure: Number; unit: Percentages
Arm/Group | <=5% Percentile | >5% - 25% Percentile | >25% - 50% Percentile | >50% - 75% Percentile | >75% - 95% Percentile | >95% Percentile | Total
Number analyzed (Participants) | 15 | 10 | 7 | 11 | 6 | 1 | 50
Percentages
  Decrease | 0.0 | 20.0 | 42.9 | 72.7 | 16.7 | 0.0 | 28.0
  No Change | 33.3 | 20.0 | 0.0 | 18.2 | 33.3 | 100.0 | 24.0
  Increase >3 to 5% | 0.0 | 0.0 | 0.0 | 0.0 | 16.7 | 0.0 | 2.0
  Increase >5 to 10% | 26.7 | 0.0 | 0.0 | 9.1 | 0.0 | 0.0 | 10.0
  Increase >10% | 40.0 | 60.0 | 57.1 | 0.0 | 33.3 | 0.0 | 36.0

6. Secondary Outcome: Growth Development - Weight at Baseline and Month 24
Description: as for outcome 4
Time Frame: Baseline, Month 24
Population: Safety Analysis Set
Measure: Number; unit: Percentages
Arm/Group | <=5% Percentile | >5% - 25% Percentile | >25% - 50% Percentile | >50% - 75% Percentile | >75% - 95% Percentile | >95% Percentile | Total
Number analyzed (Participants) | 6 | 5 | 2 | 8 | 0 | 1 | 22
Percentages
  Decrease | 0.0 | 40.0 | 100.0 | 12.5 |  | 0.0 | 22.7
  No Change | 50.0 | 0 | 0.0 | 25.0 |  | 100.0 | 27.3
  Increase >3 to 5% | 16.7 | 0 | 0.0 | 12.5 |  | 0.0 | 9.1
  Increase >5 to 10% | 16.7 | 20.0 | 0.0 | 12.5 |  | 0.0 | 13.6
  Increase >10% | 16.7 | 40.0 | 0.0 | 37.5 |  | 0.0 | 27.3

7. Secondary Outcome: Growth Development - Height at Baseline and Month 24
Description: as for outcome 4
Time Frame: Baseline, Month 24
Population: Safety Analysis Set
Measure: Number; unit: Percentages
Arm/Group | <=5% Percentile | >5% - 25% Percentile | >25% - 50% Percentile | >50% - 75% Percentile | >75% - 95% Percentile | >95% Percentile | Total
Number analyzed (Participants) | 6 | 8 | 3 | 2 | 2 | 1 | 22
Percentages
  Decrease | 0.0 | 12.5 | 33.3 | 0.0 | 0.0 | 0.0 | 9.00
  No Change | 50.0 | 12.5 | 0.0 | 0.0 | 50.0 | 100.0 | 27.3
  Increase >3 to 5% | 33.3 | 12.5 | 0.0 | 0.0 | 50.0 | 0.0 | 18.2
  Increase >5 to 10% | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 4.5
  Increase >10% | 16.7 | 62.5 | 33.3 | 100.0 | 0.0 | 0.0 | 40.9

ADVERSE EVENTS:
Time Frame: Day 1 to month 24.
Description: The incidence of AEs (including infections), by primary preferred terms sorted by system organ class were collected on Day 1 and last day with study medication plus 7 days.
Groups:
- All Patients: All patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 43/56
Other Adverse Events (participants affected / at risk) | 51/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=56)
Anaemia (Blood and lymphatic system disorders) | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Splenic lesion (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Aphthous ulcer (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Internal hernia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 3
Oesophagitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pyrexia (General disorders) | 9
Bile duct stenosis (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 2
Hepatic vein occlusion (Hepatobiliary disorders) | 1
Hepatocellular injury (Hepatobiliary disorders) | 1
Portal fibrosis (Hepatobiliary disorders) | 1
Food allergy (Immune system disorders) | 1
Transplant rejection (Immune system disorders) | 2
Adenoviral upper respiratory infection (Infections and infestations) | 1
Adenovirus infection (Infections and infestations) | 3
Alpha haemolytic streptococcal infection (Infections and infestations) | 1
Bacterial pyelonephritis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Cholangitis infective (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Diarrhoea infectious (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Enterovirus infection (Infections and infestations) | 2
Epstein-Barr viraemia (Infections and infestations) | 3
Epstein-Barr virus infection (Infections and infestations) | 2
Escherichia infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 6
Gastroenteritis adenovirus (Infections and infestations) | 1
Gastroenteritis rotavirus (Infections and infestations) | 1
Gastroenteritis sapovirus (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Mastoiditis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral viral infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Puncture site infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 2
Rhinovirus infection (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Varicella zoster virus infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 2
Complications of transplanted liver (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Transplant failure (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 1
Body temperature increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Drug level increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 5
Liver function test increased (Investigations) | 2
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Headache (Nervous system disorders) | 1
Food aversion (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=56)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 4
Ear pain (Ear and labyrinth disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 22
Mouth ulceration (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 4
Pain (General disorders) | 3
Pyrexia (General disorders) | 22
Bronchitis (Infections and infestations) | 5
Conjunctivitis (Infections and infestations) | 6
Cytomegalovirus viraemia (Infections and infestations) | 5
Diarrhoea infectious (Infections and infestations) | 3
Ear infection (Infections and infestations) | 6
Epstein-Barr viraemia (Infections and infestations) | 10
Epstein-Barr virus infection (Infections and infestations) | 7
Eye infection (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 5
Influenza (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 15
Otitis media (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 14
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 7
Hepatic enzyme increased (Investigations) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Based on DMC recommendation, enrolment was terminated and patients below 7 years were converted form study medication to local standard of care but patients were followed up until Month 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.